CLINICAL TRIAL: NCT06397209
Title: Comparative Effects of Propioceptive Neuromascular Facilitation and Neural Flossing on Balance and Gait in Diabetic Peripheral Neuropathy
Brief Title: Comparative Effects of Propioceptive Neuromascular Facilitation and Neural Flossing in Diabetic Neuropathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0275
Record Dates: First submitted 2024-04-29; First posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Diabetic Peripheral Neuropathy
Keywords: Diabetic Peripheral Neuropathy; Michigan Neuropathy Screening Instrument; Neural Flossing; Propioceptive Neuromascular facilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- proprioceptive neuromuscular facilitation (Experimental): Propioceptive neuromascular facilitation alongwith routine therapy
  Interventions: Other: Propioceptive Neuromascular facilitation
- Neural flossing (Active Comparator): Neural flossing alongwith routine therapy
  Interventions: Other: Neural Flossing

INTERVENTIONS:
Other: Propioceptive Neuromascular facilitation — Propioceptive Neuromascular Facilitation techniques will be given for 5 days/week,10 repetitions,30 minutes/day for 8 weeks
  Arms: proprioceptive neuromuscular facilitation
Other: Neural Flossing — Neural Flossing exercises will be given for 5 days/week, 3 sets of 10 repetitions in 2 minutes for 30 minutes for 8 weeks
  Arms: Neural flossing

SUMMARY:
To compare the effects of propioceptive neuromascular facilitation and neural flossing on balance and gait in diabetic peripheral neuropathy.

DETAILED DESCRIPTION:
In 2023,conducted systematic review to evaluate the effects of Tai Chi on postural control in people with PN. The meta-analysis found that Tai Chi therapy for people with PN resulted in a smaller sway area, in the double-leg stance with eyes closed test , than that observed in the control group, greater distance covered in the six-minute walking test and faster performance in the timed-up-and-go test, than the baseline. Tai chi effectively enhanced dynamic postural control in people with PN. However, no better effects on postural control from Tai Chi than from other rehabilitation approaches were observed in this study.

In 2023,compare the effects of Functional strength training Versus Neurodynamic exercises on Balance and Gait of patients with Diabetic Peripheral Neuropathy. Both Functional Strength Training Exercises and Neurodynamic Exercises were found to improve the Balance and Gait in patients with Diabetic Peripheral Neuropathy. However, the Functional Strength Training showed more significantly improvement in Balance and Gait subsequently reducing fall and fall risk injury.

As per researcher knowledge, there is no comprehensive study comparing the effects of Proprioceptive Neuromuscular Facilitation (PNF) and Neural Flossing on balance and gait in individuals with diabetic neuropathy. While both methods have been studied independently, a direct head-to-head comparison is needed. Understanding the advantages and limitations of each approach in the context of diabetic neuropathy could provide valuable insights for clinicians and researchers.

ELIGIBILITY:
Inclusion Criteria:

* Clinically Diagnosed with type I and II diabetes
* Patients 45 to 65 years of age
* The participants who scored <3 as per the Michigan Neuropathy Screening Instrument (MNSI) were included in the study.
* Able to stand and walk without assistance

Exclusion Criteria:

* Patients have other neurological or orthopedic impairments (such as stroke,cerebral palsy, poliomyelitis, rheumatoid arthritis, prosthesis, or moderate or severe osteoarthritis)
* Major vascular complications (venous or arterial ulcers).
* Severe retinopathy
* Severe nephropathy that causes edema or requires haemodialysis

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-12-23 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Berg balance scale | 8th week
  The BBS was developed to assess the balance among elderly people with impairment in balance function by measuring the performance of functional tasks. It is a 14-item scale designed to measure the balance of the older adults in a clinical setting, and the maximum score of the scale is 56.The score between the ranges of 41-56 is considered to below risk fall, whereas 21-40 and 0-20 are considered to be medium risk fall and high risk fall, respectively.
Dynamic Gait Index | 8th week
  DGI assesses a person's ability to modify balance while walking in the presence of external demands. DGI is performed with a marked distance of 20 feet either with or without assistive devices. The scoring is based on a 4- point scale, and the highest possible score is 24 points. DGI score between 21 and 24 depicts safe ambulatory, whereas score of <21 is predictive of falls.

CONTACTS AND LOCATIONS:
Overall Officials: Sana Akram, DPT, Principal Investigator — Riphah International University (Lahore)
Locations (1):
- Dhillon Surgical Hospital, Burewala, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mirek E, Filip M, Banaszkiewicz K, Rudzinska M, Szymura J, Pasiut S, Stozek J, Szczudlik A. The effects of physiotherapy with PNF concept on gait and balance of patients with Huntington's disease - pilot study. Neurol Neurochir Pol. 2015;49(6):354-7. doi: 10.1016/j.pjnns.2015.09.002. Epub 2015 Sep 15. PMID 26652868
- [Background] Khan KS, Andersen H. The Impact of Diabetic Neuropathy on Activities of Daily Living, Postural Balance and Risk of Falls - A Systematic Review. J Diabetes Sci Technol. 2022 Mar;16(2):289-294. doi: 10.1177/1932296821997921. Epub 2021 Mar 14. PMID 33719603
- [Background] Boyd BS, Nee RJ, Smoot B. Safety of lower extremity neurodynamic exercises in adults with diabetes mellitus: a feasibility study. J Man Manip Ther. 2017 Feb;25(1):30-38. doi: 10.1080/10669817.2016.1180772. Epub 2016 Jun 17. PMID 28855790
- [Background] Kluding PM, Bareiss SK, Hastings M, Marcus RL, Sinacore DR, Mueller MJ. Physical Training and Activity in People With Diabetic Peripheral Neuropathy: Paradigm Shift. Phys Ther. 2017 Jan 1;97(1):31-43. doi: 10.2522/ptj.20160124. PMID 27445060
- [Background] Metsker O, Magoev K, Yakovlev A, Yanishevskiy S, Kopanitsa G, Kovalchuk S, Krzhizhanovskaya VV. Identification of risk factors for patients with diabetes: diabetic polyneuropathy case study. BMC Med Inform Decis Mak. 2020 Aug 24;20(1):201. doi: 10.1186/s12911-020-01215-w. PMID 32831065
- [Background] Mao W, Wang T, Sun M, Zhang F, Li L. Effects of Tai Chi on Postural Control in People with Peripheral Neuropathy: A Systematic Review with Meta-Analysis. Healthcare (Basel). 2023 May 26;11(11):1559. doi: 10.3390/healthcare11111559. PMID 37297699
- [Background] Ernandes RC, Brech GC, Luna NMS, Bega A, GuimarAes DS, Bocalini DS, Scherrer G, Greve JMD, Leme LEG, Alonso AC. IMPACT OF DIABETIC NEUROPATHY ON QUALITY OF LIFE AND POSTURAL BALANCE IN BRAZILIAN OLDER ADULTS. Acta Ortop Bras. 2020 Nov-Dec;28(6):275-279. doi: 10.1590/1413-785220202806234529. PMID 33328782
- [Background] Jamal A, Ahmad I, Ahamed N, Azharuddin M, Alam F, Hussain ME. Whole body vibration showed beneficial effect on pain, balance measures and quality of life in painful diabetic peripheral neuropathy: a randomized controlled trial. J Diabetes Metab Disord. 2019 Dec 21;19(1):61-69. doi: 10.1007/s40200-019-00476-1. eCollection 2020 Jun. PMID 32550157
- [Background] Sartor CD, Watari R, Passaro AC, Picon AP, Hasue RH, Sacco IC. Effects of a combined strengthening, stretching and functional training program versus usual-care on gait biomechanics and foot function for diabetic neuropathy: a randomized controlled trial. BMC Musculoskelet Disord. 2012 Mar 19;13:36. doi: 10.1186/1471-2474-13-36. PMID 22429765
- [Background] Barbosa M, Saavedra A, Severo M, Maier C, Carvalho D. Validation and Reliability of the Portuguese Version of the Michigan Neuropathy Screening Instrument. Pain Pract. 2017 Apr;17(4):514-521. doi: 10.1111/papr.12479. Epub 2016 Aug 19. PMID 27538385
- [Background] Godi M, Franchignoni F, Caligari M, Giordano A, Turcato AM, Nardone A. Comparison of reliability, validity, and responsiveness of the mini-BESTest and Berg Balance Scale in patients with balance disorders. Phys Ther. 2013 Feb;93(2):158-67. doi: 10.2522/ptj.20120171. Epub 2012 Sep 27. PMID 23023812
- [Background] Jonsdottir J, Cattaneo D. Reliability and validity of the dynamic gait index in persons with chronic stroke. Arch Phys Med Rehabil. 2007 Nov;88(11):1410-5. doi: 10.1016/j.apmr.2007.08.109. PMID 17964880
- [Background] Sharma S, Kalia V. Effect of tibial nerve mobilization on balance & gait functions in subjects with subclinical diabetic neuropathy: A randomized clinical trial. J Diabetes Metab Disord. 2023 Aug 16;22(2):1283-1290. doi: 10.1007/s40200-023-01246-w. eCollection 2023 Dec. PMID 37975109